CLINICAL TRIAL: NCT01908738
Title: Effectiveness of Paracervical Block Versus Lidocaine Spray During Endometrial Biopsy Under Oral Analgesic Drugs; A Randomized Controlled Trial
Brief Title: Effectiveness of Paracervical Block Versus Lidocaine Spray During Endometrial Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Akarawit Jitchanwichai, faculty of medicine obstertic and gynecology, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 56-244-12-4-2
Record Dates: First submitted 2013-07-18; First posted 2013-07-26 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2014-03

CONDITIONS: Endometrial Biopsy; Abnormal Uterine Bleeding
Keywords: Endometrial biopsy; paracervical block; Lidocaine spray; women; abnormal uterine bleeding
MeSH Terms: conditions — Metrorrhagia | interventions — Anesthesia, Obstetrical

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- paracervical block with 1%lidocaine and 0.9%NSS spray(placebo) (Experimental): first groups receive paracervical block with 1%lidocaine and 0.9%NSS spray(placebo)
  Interventions: Drug: paracervical block with 1%lidocaine
- 10%lidocaine spray and paracervical block with 0.9%NSS (Experimental): the second groups receive 10%lidocaine spray and paracervical block with 0.9%NSS(placebo)
  Interventions: Drug: 10%lidocaine spray
- receive placebo both paracervical block and spray (Placebo Comparator): the third groups receive placebo both paracervical block and spray
  Interventions: Drug: paracervical block with 1%lidocaine; Drug: 10%lidocaine spray

INTERVENTIONS:
Drug: paracervical block with 1%lidocaine — To determine effectiveness of paracervical block, lidocaine spray and only oral analgesic drugs for pain relief during endometrial biopsy.
  Pain score(NRS) immediately after procedure and 15 minutes Group 1(1%Lidocaine) Group 2(10%Lidocaine spray) Control group(Placebo) Pain score immediately Pain score 15 minutes
  Arms: paracervical block with 1%lidocaine and 0.9%NSS spray(placebo); receive placebo both paracervical block and spray
Drug: 10%lidocaine spray
  Arms: 10%lidocaine spray and paracervical block with 0.9%NSS; receive placebo both paracervical block and spray

SUMMARY:
The purpose of this study to determine effectiveness of paracervical block, lidocaine spray and only oral analgesic drugs for pain relief during endometrial biopsy.

DETAILED DESCRIPTION:
Participants : This study was conducted prospectively at the outpatient clinic, Department of Obstetrics and Gynecology, Songklanagarind Hospital.

Inclusion criteria : The women who had abnormal uterine bleeding and indication for endometrial biopsy were enrolled.

Exclusion criteria : included 1) contraindications to NSAID or Lidocaine - known sensitivity to these drugs; 2) pregnancy; 3) genital tract infection; 4) coagulation disorder; and 5) unstable vital signs.

Sample size calculation : Sample size was calculated by assuming the different mean pain score of each groups performing the endometrial biopsy to be 1. To evidence this difference with a power of 80% and a 5% level of significance, a need was calculated with 36 women in each group and for total was 108 women.

Z α/2 = Type I error(alpha error) α = 0.05 >> 1.96 Z β = Type II error(beta error) β = 0.2 >> 0.84

* Variance of mean pain score between procedure and post procedure 15 minutes = 1.5 µ0 = Mean pain score in group 1 µ1 = Mean pain score in group 2 µ0 - µ1 = Different of mean pain score in between each groups = 1 **N = 2(1.5)2(1.96 + 0.84)2/(1)2 = 35.3 N = 36 per group

Study procedures :

1. Explain the steps of the procedure to the patient and counseling regarding rational and risks/benefits. Obtain consent for the procedure. Perform bimanual exam to determine uterine size and position.
2. After signing a written informed consent, the women were randomly allocated to 3 groups. All women will receive Acetaminophen 500 mg and Ibuprofen 400 mg before procedure 30 minutes.

   The first groups receive paracervical block with 1%lidocaine and 0.9%NSS spray(placebo), the second groups receive 10%lidocaine spray and paracervical block with 0.9%NSS(placebo) and the third groups receive placebo both paracervical block and spray. Both women and researcher associate were blinded to group allocation. The 1%lidocaine, 10%lidocaine spray and both placebos were prepared in sequentially numbered sealed opaque envelops according to the table of random numbers by an independent pharmacist.
3. The time that start oral medication and vital signs before starting procedure were recorded.
4. Starting procedure by using largest appropriate speculum for maximum cervical exposure. Cleanse the cervix with povidone iodine. Then administer paracervical block by using local anesthetic drug 5 ml. injects at cervical area 3 and 9 O'clock, depth 0.5-1 cm., 2.5 ml. each sides. After that use anesthetic spray sprays at cervix for 1 times and wait for 3 minutes.
5. Endometrial biopsy was performed by using a 3-mm EndosamplerTM (MedGyn EndosamplerTM, MedGyn Product Inc, IL, USA). If insertion of EndosamplerTM failed, a tenaculum was applied to the anterior cervix to help for stabilization and counter-traction.
6. After get the endometrial tissue sample, remove all equipments, checked and stopped bleeding. And record vital signs after finish the procedure.
7. The form contained a visual analog scale for women to report their responses of pain at immediately after procedure and after that 15 minutes by using Numerical Rating Scale(NRS) were recorded.
8. The women were assessed for adverse side effects or complications of procedure e.g. such as dizziness, nausea, vomiting, pelvic pain or others.
9. Follow up appointment the women for pathological report result at PSU hospital and consider further management.

Expected outcomes :

To determine effectiveness of paracervical block, lidocaine spray and only oral analgesic drugs for pain relief during endometrial biopsy.

Table. Pain score(NRS) immediately after procedure and 15 minutes Group 1(1%Lidocaine) Group 2(10%Lidocaine spray) Control group(Placebo) Pain score immediately Pain score 15 minutes A secondary goal of this study was to determine the adverse effects of these methods(such as dizziness, nausea, vomiting, pelvic pain, bleeding).

Data analysis :

Data are presented as median (range) for quantitative variables and frequency for qualitative variables. Comparison between both groups was made by using the Chi-square test, Fisher's exact test and Mann-Whitney U test where appropriate with p<0.05 considered statistically significant. Statistical analysis was performed with the SPSS 17.0 package program (Statistical Package for Social Science; SPSS Inc., Chicago, IL, USA).

Ethical consideration :

* Inform consent will be obtained before study procedure.
* The study will not detrimental patients or treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* abnormal uterine bleeding women
* indicated for endometrial biopsy

Exclusion Criteria:

1. contraindications to NSAID or Lidocaine - known sensitivity to these drugs
2. pregnancy
3. genital tract infection
4. coagulation disorder
5. unstable vital signs.

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Effectiveness of paracervical block VS Lidocaine spray during endometrial biopsy ; A randomized controlled trial | up to 12 months
  measurement outcome by record Pain score(NRS)[Numberical rating scale 0-10] immediately after procedure and 15 minutes after procedure in all groups Group 1(1%Lidocaine) Group 2(10%Lidocaine spray) Group 3 Control group(Placebo) Pain score immediately and Pain score 15 minutes were compared between group by using statistic analysis to indentify the significant of decreasing Pain score for pain relief during endometrial biopsy.
  And after that the result will used to determine effectiveness of each groups[ paracervical block, lidocaine spray and only oral analgesic drugs.

SECONDARY OUTCOMES:
adverse effects of paracervical block versus lidocaine spray | up to 12 months
  A secondary goal of this study was to determine the adverse effects of these methods(such as dizziness, nausea, vomiting, pelvic pain, bleeding) by recording the adverse effects outcome of each groups and report the result.

CONTACTS AND LOCATIONS:
Locations (1):
- Akarawit Jitchanwichai, Songkhla, Hatyai, Thailand